CLINICAL TRIAL: NCT00472732
Title: Assessing Neural Mechanisms of Injury in Inborn Errors of Urea Metabolism Using Structural MRI, Functional MRI, and Magnetic Resonance Spectroscopy
Brief Title: Neurologic Injuries in Adults With Urea Cycle Disorders
Status: Completed | Type: Observational
Sponsor: Andrea Gropman (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); Rare Diseases Clinical Research Network (Network); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Andrea Gropman, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: RDCRN 5104; U54RR019453 (NIH)
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-05

CONDITIONS: Brain Diseases, Metabolic, Inborn; Urea Cycle Disorder; Ornithine Transcarbamylase Deficiency
Keywords: UCD; OTCD; Ammonia; Urea Metabolism; Inborn Errors
MeSH Terms: conditions — Brain Diseases, Metabolic, Inborn; Urea Cycle Disorders, Inborn; Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Female carriers of ornithine transcarbamylase deficiency (OTCD) or males with late onset presentation of OTCD
- 2: Healthy males or females without known medical or metabolic disorder (control group)

SUMMARY:
Urea cycle disorders (UCDs) are a group of rare inherited metabolism disorders. The purpose of this study is to evaluate how UCD-related neurologic injuries affect adults with one of the most common types of UCD.

DETAILED DESCRIPTION:
UCDs are a group of rare genetic diseases that affect how protein is broken down in the body. The cause of UCDs is a deficiency in one of eight enzymes responsible for removing ammonia, a waste product of protein metabolism, from the bloodstream. Normally, ammonia is converted into urea and then removed from the body in the form of urine. However, in people with UCDs, ammonia accumulates unchecked and is not removed from the body. Toxic levels of ammonia can build up and cause irreversible neurologic damage that can affect metabolism, cognition, sensation, and movement. This study will focus on the most common enzyme disorder among UCDs, ornithine transcarbamylase deficiency (OTCD), a disorder inherited from mothers. Using different types of magnetic resonance imaging (MRI), this study will evaluate how UCD-related neurologic injuries affect metabolism, cognition, sensation, and movement in adults with OTCD.

Participants in this study will attend an initial study visit that will include a review of medical history, current symptoms, impairments, and diet history; urine and blood collection; a physical exam; a full neurological exam; and cognitive and motor testing. During this visit, participants will undergo imaging studies and additional cognitive and motor testing over a 2- to 3-day period. This will include standard MRI studies and four sessions consisting of functional MRI (fMRI), diffusion tensor imaging, and 1H magnetic resonance spectroscopy. For the fMRI study, participants perform various motor and behavioral tasks while in the imaging scanner. Magnetic resonance spectroscopy (MRS) is used to study and evaluate the chemical makeup of specific brain areas. Diffusion tensor imaging is used to assess myelination of major brain pathways and their alteration in disease states. This study will involve one-time participation. There will be no follow-up visits for this study.

ELIGIBILITY:
Inclusion Criteria for Participants with OTCD:

* Diagnosis of OTCD or heterozygote state of OTCD by metabolic or molecular means. Female participants must be clinically stable and heterozygous for OTCD. Male participants must be hemizygous for late onset OTCD.

Inclusion Criteria for Healthy Controls:

* No known medical or metabolic disorder

Inclusion Criteria for All Participants:

* IQ of at least 80
* Willing to travel to study site
* English-speaking
* Age between 18 and 60 years

Exclusion Criteria for All Participants:

* Currently being treated for an acute illness
* History of neuropsychiatric drug use
* Unable to undergo MRI scanning without being sedated
* Unable to participate in neurocognitive and/or motor testing
* Metal device in body that might interfere with MRI scanning
* Pregnancy or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female carriers of ornithine transcarbamylase deficiency (OTCD) or males with late onset presentation of OTCD
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2007-03; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Gropman, MD, Study Chair — Children's National Research Institute
Locations (2):
- United States (2):
  - George Washington University School of Medicine, Washington D.C., District of Columbia
  - Georgetown University, Washington D.C., District of Columbia

REFERENCES:
- [Background] Gyato K, Wray J, Huang ZJ, Yudkoff M, Batshaw ML. Metabolic and neuropsychological phenotype in women heterozygous for ornithine transcarbamylase deficiency. Ann Neurol. 2004 Jan;55(1):80-6. doi: 10.1002/ana.10794. PMID 14705115
- [Background] Kurihara A, Takanashi Ji, Tomita M, Kobayashi K, Ogawa A, Kanazawa M, Yamamoto S, Kohno Y. Magnetic resonance imaging in late-onset ornithine transcarbamylase deficiency. Brain Dev. 2003 Jan;25(1):40-4. doi: 10.1016/s0387-7604(02)00153-5. PMID 12536032
- [Background] McCullough BA, Yudkoff M, Batshaw ML, Wilson JM, Raper SE, Tuchman M. Genotype spectrum of ornithine transcarbamylase deficiency: correlation with the clinical and biochemical phenotype. Am J Med Genet. 2000 Aug 14;93(4):313-9. doi: 10.1002/1096-8628(20000814)93:43.0.co;2-m. PMID 10946359

RESULTS

PARTICIPANT FLOW:
Groups:
- Female Carriers of Ornithine Transcarbamylase Deficiency (OTCD: Female carriers of ornithine transcarbamylase deficiency (OTCD) or males with late onset presentation of OTCD
- Healthy Males or Females Without Known Medical or Metabolic di: Healthy males or females without known medical or metabolic disorder (control group)
Period: Overall Study
Arm/Group | Female Carriers of Ornithine Transcarbamylase Deficiency (OTCD | Healthy Males or Females Without Known Medical or Metabolic di
Started | 24 | 22
Completed | 24 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Half of the subjects were affected and half were normal controls age 18-60
Groups:
- Total: Total of all reporting groups
Arm/Group | Female Carriers of Ornithine Transcarbamylase Deficiency (OTCD | Healthy Males or Females Without Known Medical or Metabolic di | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Customized [Mean (Full Range); unit: years]
  Age | 32.55 [18 to 58] | 32.38 [18 to 59] | 32.46 [18 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 23 | 21 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 5 | 5
  White | 23 | 15 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 22 | 46

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Glutamine and Myoinositol by MRS
Description: Concentration based on area under curve on 1H MRS and quantitated by LCModel. A metabolite's tissue concentration is related to the integrated amplitude of the MRS signal it produces. Integrated amplitude is the area under the MRS signal curve. While MRS signals are usually acquired in the time domain as free induction decays or echoes, they are usually viewed and analyzed in the frequency domain. The frequency domain representation is derived from the acquired time domain data by the Fourier Transform. The protocol we use selects 257 averages. This means, 257 free induction decays. The machine summates the data at each time point to generate one value for the area under the curve. Therefore, we don't have the measurement at each time point.
  Furthermore, we measured voxels in two different brain areas containing different kinds of brain matter: one voxel was located in posterior cingulate gray matter (PCGM) and the other in parietal white matter (PWM).
Time Frame: one time measurement at study baseline
Measure: Mean (Standard Deviation); unit: mM
Groups:
- OTCD Patients: Female carriers of ornithine transcarbamylase deficiency (OTCD) or males with late onset presentation of OTCD
- Healthy Controls: Healthy males or females without known medical or metabolic disorder (control group)
Arm/Group | OTCD Patients | Healthy Controls
Number analyzed (Participants) | 24 | 22
mM
  Glutamine in PCGM | 4.97 (2.08) | 3.66 (1.36)
  Myoinositol in PCGM | 3.78 (0.82) | 4.50 (0.43)
  Glutamine in PWM | 2.13 (1.22) | 1.09 (0.75)
  Myoinositol in PWM | 2.27 (0.77) | 2.86 (0.38)
Statistical Analysis 1: Comparison: OTCD Patients vs Healthy Controls; The null hypothesis predicted that the concentration of myoinositol in posterior cingulate gray matter will be the same in OTCD patients as in controls; Test type: Superiority or Other; p = 0.003, t-test, 2 sided — The Bonferroni-corrected a priori p-value was 0.007 (a priori alpha=0.05/number of tests=7)
Statistical Analysis 2: Comparison: OTCD Patients vs Healthy Controls; The null hypothesis predicted that the concentration of myoinositol in parietal white matter will be the same in OTCD patients as in controls; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The Bonferroni-corrected a priori p-value was 0.007 (a priori alpha=0.05/number of tests=7)
Statistical Analysis 3: Comparison: OTCD Patients vs Healthy Controls; The null hypothesis predicted that the concentration of glutamine in posterior cingulate gray matter would be the same for OTCD patients as for controls; Test type: Superiority or Other; p = 0.001, t-test, 2 sided — The Bonferroni-corrected a priori p-value was 0.007 (a priori alpha=0.05/number of tests=7)
Statistical Analysis 4: Comparison: OTCD Patients vs Healthy Controls; The null hypothesis predicted that the concentration of glutamine in parietal white matter would be the same for OTCD patients as for controls; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The Bonferroni-corrected a priori p-value was 0.007 (a priori alpha=0.05/number of tests=7)

2. Primary Outcome: Functional MRI Activation in N-Back Tast
Description: Measure of blood oxygen level dependent (BOLD) signal of OTCD patients and healthy controls during an N-Back task comparing 2-back and 1-back conditions. This contrast was created for each participant using SPM and then entered into a group analysis in which we compare percent signal change between groups. Therefore, we never see BOLD signal change at the individual level, which is why we never see "scores" or numbers at the individual level and we cannot calculate a measure of dispersion for this data.
Time Frame: one time measurement at study baseline
Population: Five OTCD patients and one healthy control were excluded due to excessive head motion.
Measure: Number; unit: percent signal change
Arm/Group | OTCD Patients | Healthy Controls
Number analyzed (Participants) | 19 | 21
percent signal change
  Dorsolateral prefrontal cortex (BA 10) | 0.21 | 0.04
  Dorsolateral prefrontal cortex (BA 46) | 0.22 | 0.15
  Anterior cingulate cortex (BA 32) | 0.515 | 0.28
Statistical Analysis 1: Comparison: OTCD Patients vs Healthy Controls; Two-way between-group t-tests restricted to the prefrontal cortex were performed to compare activation during for the 2-Back> 1-Back contrast between OTCD patients and controls; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — This p-value is adjusted for family wise error rate correction

3. Primary Outcome: Fractional Anisotropy
Description: Measure of white matter integrity in OTCD Patients and Controls in frontal white matter. Fractional anisotropy values fall on a scale of 0 to 1, with 0 meaning that the diffusion of water is isotropic and unrestricted, or equally restricted, in all directions and with 1 meaning that diffusion occurs along only one axis and is fully restricted along all other directions. Scores closer to 1 are associated with intact white matter while scores closer to 0 are associated with white matter damage.
Time Frame: one time measurement at study baseline
Population: Five OTCD Patients and four healthy controls were excluded due to excessive head motion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OTCD Patients | Healthy Controls
Number analyzed (Participants) | 19 | 18
units on a scale | 0.247 (0.016) | 0.274 (0.015)
Statistical Analysis 1: Comparison: OTCD Patients vs Healthy Controls; The null hypothesis predicted that fractional anisotropy, a marker of white matter integrity, would be the same for OTCD patients as for controls; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Entire study
Arm/Group | OTCD Patients | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 0/24 | 0/22

LIMITATIONS AND CAVEATS:
This study examined the neurobiological differences between OTCD patients and controls. This was, however, not a clinical trial, since participants received no form of drug therapy or treatment as part of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No